CLINICAL TRIAL: NCT00607152
Title: A Multi-center, Randomized, Open-label, Active-controlled Clinical Trial to Evaluate the Efficacy and Safety of Rasburicase (Fasturtec®) in the Prevention and Treatment of Hyperuricemia in Patients With Hematological Malignancies
Brief Title: Rasburicase (Fasturtec) Registration Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: the patient enrollment is too difficult
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RASBU_L_00351
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Hyperuricemia
MeSH Terms: conditions — Hyperuricemia | interventions — rasburicase; Allopurinol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): IV infusion at a dose level of 0.20mg/kg per day
  Interventions: Drug: Rasburicase
- 2 (Active Comparator): 100mg tablets, administered orally, according to standard medical practice
  Interventions: Drug: Allopurinol

INTERVENTIONS:
Drug: Rasburicase — 0.20mg/kg per day IV
  Arms: 1
Drug: Allopurinol — 100mg tablets
  Arms: 2

SUMMARY:
Primary:

To compare the efficacy of Rasburicase versus allopurinol in controlling tumor lysis-related hyperuricemia in Chinese patients with leukemia or lymphoma.

Secondary:

To compare the efficacy and safety of Rasburicase versus allopurinol in Chinese patients stratified according to disease (leukemia or lymphoma ).

ELIGIBILITY:
Inclusion Criteria:

* At high risk of malignancy and/or chemotherapy-induced hyperuricemia
* Performance status less than 3 on ECOG scale or more than 30% KPS scale
* Uric acid concentrations ≥ 8.0mg/dL
* Suffering from non-Hodgkin's lymphoma Stage more than III, or acute lymphoblastic leukemia with peripheral with blood cell count more than 25,000/mm3, or any lymphoma or leukemia

Exclusion Criteria:

* Treatment with an investigational drug at any time during the 14-day study period (except for agents that are permitted by the Sponsor)
* Pregnancy or lactation
* Prior treatment with Uricozyme or Rasburicase
* Scheduled to receive asparaginase either 24 hours after the first dose of rasburicase
* Treatment with Allopurinol within the seven days preceding study Day 1
* History of significant atopic allergy problems or documented history of asthma
* History of severe reaction to allopurinol
* Known history of glucose-6-phosphate dehydrogenase deficiency.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Mean plasma uric acid AUC0-96 | 0hour, 4hour, 12 hour and q12h thereafter
Median duration of therapy until control of plasma uric acid values to <8.0 mg/dL (only in patients hyperuricemic immediately prior to dosing) | From administration of drug up to end of study
Biochemistry, hematology, vital signs, physical examination, and adverse events | From administration of drug up to end of study
Proportion of patients developing hypertension requiring therapy | From administration of drug up to end of study
Assays for circulating antibodies | From administration of drug up to end of study

SECONDARY OUTCOMES:
Percentage reduction of plasma uric acid concentrations at T4h | From administration of drug up to end of study
Mean plasma uric acid concentrations | At various timepoints
Median duration of therapy until control of plasma uric acid values to <8.0 mg/dL | From administration of drug up to end of study

CONTACTS AND LOCATIONS:
Overall Officials: Jing Fu, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China